CLINICAL TRIAL: NCT04135196
Title: A Prospective Study of Human Bone Adaptation Using a Novel in Vivo Loading Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Worcester Polytechnic Institute (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13-111
Record Dates: First submitted 2019-07-19; First posted 2019-10-22 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-01

CONDITIONS: Bone Loss
Keywords: bone; adaptation; mechanical stimuli; women; peak bone mass
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: all data were blinded for analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low Magnitude (Experimental): voluntary forearm compression by leaning onto the palm of the hand with low target strain
  Interventions: Other: voluntary forearm loading task
- High Magnitude (Experimental): voluntary forearm compression by leaning onto the palm of the hand with high target strain
  Interventions: Other: voluntary forearm loading task
- Low Rate (Experimental): voluntary forearm compression by leaning onto the palm of the hand with low strain rate (task performed "slowly and evenly")
  Interventions: Other: voluntary forearm loading task
- High Rate (Experimental): voluntary forearm compression by leaning onto the palm of the hand with high strain rate (task performed "as quickly as possible, with a bump")
  Interventions: Other: voluntary forearm loading task
- Control (No Intervention): observation only

INTERVENTIONS:
Other: voluntary forearm loading task — voluntary task, consisting of leaning onto the palm of the hand until a target force is reached. Each loading bout consists of 100 loading cycles, which takes approximately 2 minutes to complete. The task is performed 4 times per week during the intervention period.
  Arms: High Magnitude; High Rate; Low Magnitude; Low Rate

SUMMARY:
The purpose of this study is to understand how different types of mechanical forces can influence bone adaptation (and make bones stronger, potentially). Forces acting on bones cause mechanical strain. In small animals, strain magnitude and rate have been shown to stimulate bone adaptation. This study is designed to test the degree to which strain magnitude and rate govern bone adaptation in healthy adult women.

DETAILED DESCRIPTION:
The study consists of three Aims:

Aim 1: compare the effect on bone structure of mechanical signals with low strain magnitude, high strain magnitude, and control groups over a 12-month prospective period.

Aim 2. Compare the effect on bone structure of mechanical signals with low strain rate, high strain rate, and control groups over a 12-month prospective period.

Aim 3: Examine the effect of withdrawing mechanical signals, by measuring bone structure during the 12 months after the intervention is withdrawn.

The intervention is a voluntary forearm compression task, consisting of leaning onto the palm of the hand to produce a target force.

The primary outcome measure is change in distal radius bone mineral content (BMC).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21-40
* Body Mass Index [18-29]
* 9-14 menstrual cycles/year
* Dual energy X-ray Absorptiometry total radius bone mineral density (BMD) T-score [-2.5-+1]
* Free of endocrinopathies
* No known thyroid, vitamin D, or calcium abnormalities

Exclusion Criteria:

* Fracture to wrist <5 years ago
* Wrist Arthritis
* Injury to the non-dominant elbow or shoulder <5 years ago
* Diabetes
* Severe disabling conditions
* Cancer <5 years ago
* Metabolic bone disease
* Androgen, estrogen, progesterone, calcitonin, Selective Estrogen Receptor Modulators, Parathyroid hormone, gonadotropin-releasing hormone or analogs used <6 months ago
* Corticosteroids <3 months ago
* Bisphosphonates or fluoride <3 years ago
* Cardiovascular/pulmonary disease
* Uncontrolled hypertension
* Regular Tobacco use
* Marijuana use >1 time/week
* Alcohol >4 drinks/day
* Pregnancy or lactation <2 years ago
* Plan to become pregnant or donate eggs within 1 year
* Depot medroxyprogesterone acetate contraceptive <6 months ago
* Current participation in upper extremity loading sports (gymnastics, tennis, softball, hockey) >2 times/month
* Low calcium intake (avoiding dairy products without taking calcium supplement)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2019-07-19 (Actual)

REFERENCES:
- [Result] Mancuso ME, Johnson JE, Ahmed SS, Butler TA, Troy KL. Distal radius microstructure and finite element bone strain are related to site-specific mechanical loading and areal bone mineral density in premenopausal women. Bone Rep. 2018 Apr 14;8:187-194. doi: 10.1016/j.bonr.2018.04.001. eCollection 2018 Jun. PMID 29963602
- [Result] Troy KL, Mancuso ME, Johnson JE, Wu Z, Schnitzer TJ, Butler TA. Bone Adaptation in Adult Women Is Related to Loading Dose: A 12-Month Randomized Controlled Trial. J Bone Miner Res. 2020 Jul;35(7):1300-1312. doi: 10.1002/jbmr.3999. Epub 2020 Mar 30. PMID 32154945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2013-June 2017 All participants were recruited at a single site (Worcester Polytechnic Institute) and the surrounding community via social media, posters, email newsletters, and word of mouth at nearby universities, hospitals, and community events.
Period: Overall Study
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Started | 21 | 24 | 21 | 20 | 16
Completed | 13 (13 participants analyzed at 12 months 15 participants analyzed at interim timepoints) | 17 (17 participants analyzed at 12 months 21 participants analyzed at interim timepoints) | 12 (12 participants analyzed at 12 months 15 participants analyzed at interim timepoints) | 11 (11 participants analyzed at 12 months 11 participants analyzed at interim time points) | 14 (13 participants analyzed at 12 months (data not available for n=1) 15 participants analyzed at interim timepoints)
Not Completed | 8 | 7 | 9 | 9 | 2
Not completed — Lost to Follow-up | 8 | 7 | 8 | 9 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control | Total
Number analyzed (Participants) | 21 | 24 | 21 | 20 | 16 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (5.5) | 29.3 (6.3) | 27.2 (5.1) | 27.1 (5.4) | 28.2 (5.3) | 28.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 21 | 20 | 16 | 102
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 1 | 2 | 2 | 12
  Not Hispanic or Latino | 19 | 18 | 20 | 18 | 14 | 89
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 4 | 3 | 0 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 16 | 17 | 16 | 14 | 13 | 76
  More than one race | 1 | 2 | 1 | 1 | 2 | 7
  Unknown or Not Reported | 1 | 3 | 0 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 21 | 20 | 16 | 102
Height [Mean (Standard Deviation); unit: cm] | 165.8 (6.1) | 161.9 (6.1) | 165.0 (6.2) | 164.9 (5.7) | 167.3 (7.6) | 164.8 (6.4)
Body Mass [Mean (Standard Deviation); unit: kg] | 65.2 (8.8) | 61.0 (5.9) | 65.4 (9.8) | 65.4 (10) | 65.0 (8.9) | 64.3 (8.7)
Serum Vitamin D [Mean (Standard Deviation); unit: ng/mL] — circulating levels of 25-hydroxyvitamin D
  ng/mL | 33.7 (9.9) | 31.5 (8.9) | 31.1 (12.2) | 29.1 (7.8) | 33.2 (7.5) | 31.7 (9.5)
Total Forearm aBMD [Mean (Standard Deviation); unit: g/cm^2] — areal bone mineral density (BMD) in the Total region for the standard Forearm (Left or Right, non-dominant arm scanned) Analysis Protocol for the Hologic Discovery C densitometer.
  g/cm^2 | 0.586 (0.04) | 0.568 (0.03) | 0.576 (0.04) | 0.569 (0.04) | 0.570 (0.04) | 0.574 (0.04)
DXA Total Forearm T-score [Mean (Standard Deviation); unit: t-score] — Dual energy x-ray absorptiometry (DXA) total forearm t-score. This is the forearm bone mineral density, expressed in numbers of standard deviations away from the average healthy young adult value. A t-score of 0 is equal to the mean. Scores less than 0 indicate lower bone density than a race and gender matched young healthy adult population and scores greater than 0 indicate higher bone density than a race and gender matched young healthy adult population.
  t-score | 0.138 (0.76) | -0.187 (0.63) | 0.138 (0.76) | -0.175 (0.74) | -0.162 (0.67) | -0.087 (0.70)
Ultradistal iBMC [Mean (Standard Deviation); unit: g] — ultradistal integral bone mineral content measured using quantitative analysis of clinical resolution computed tomography (CT) scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for the group of participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g
    All Enrolled Participants | 0.940 (0.179) | 0.886 (0.149) | 0.894 (0.141) | 0.844 (0.155) | 0.883 (0.116) | 0.890 (0.151)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.997 (0.143) | 0.849 (0.134) | 0.926 (0.160) | 0.875 (0.140) | 0.898 (0.124) | 0.906 (0.145)
Ultradistal cBMC [Mean (Standard Deviation); unit: g] — ultradistal cortical bone mineral content measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g
    All Enrolled Participants | 0.432 (0.163) | 0.380 (0.123) | 0.369 (0.109) | 0.354 (0.104) | 0.356 (0.077) | 0.380 (0.122)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.457 (0.177) | 0.351 (0.117) | 0.377 (0.132) | 0.369 (0.104) | 0.369 (0.076) | 0.383 (0.128)
Ultradistal ecBMC [Mean (Standard Deviation); unit: g] — ultradistal endocortical bone mineral content measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g
    All Enrolled Participants | 0.692 (0.226) | 0.607 (0.181) | 0.617 (0.163) | 0.564 (0.171) | 0.597 (0.127) | 0.617 (0.180)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.745 (0.211) | 0.556 (0.149) | 0.644 (0.195) | 0.596 (0.172) | 0.613 (0.135) | 0.627 (0.180)
Ultradistal tBMC [Mean (Standard Deviation); unit: g] — ultradistal trabecular bone mineral content measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g
    All Enrolled Participants | 0.182 (0.061) | 0.177 (0.053) | 0.181 (0.053) | 0.158 (0.061) | 0.179 (0.052) | 0.175 (0.056)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.201 (0.039) | 0.166 (0.048) | 0.196 (0.062) | 0.170 (0.047) | 0.184 (0.057) | 0.182 (0.051)
Ultradistal iBV [Mean (Standard Deviation); unit: cm^3] — ultradistal integral bone volume measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  cm^3
    All Enrolled Participants | 3.88 (0.44) | 3.73 (0.34) | 3.78 (0.45) | 3.72 (0.53) | 3.79 (0.37) | 3.78 (0.43)
    Subset of Participants who were also Analyzed at Follow-up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-up (12 months) | 4.02 (0.39) | 3.70 (0.34) | 3.88 (0.38) | 3.77 (0.56) | 3.85 (0.28) | 3.84 (0.40)
Ultradistal cBV [Mean (Standard Deviation); unit: cm^3] — ultradistal cortical bone volume measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  cm^3
    All Enrolled Participants | 0.88 (0.26) | 0.80 (0.22) | 0.79 (0.20) | 0.74 (0.20) | 0.76 (0.15) | 0.79 (0.21)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.92 (0.26) | 0.74 (0.20) | 0.81 (0.25) | 0.78 (0.21) | 0.78 (0.14) | 0.80 (0.22)
Ultradistal ecBV [Mean (Standard Deviation); unit: cm^3] — ultradistal endocortical bone volume measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  cm^3
    All Enrolled Participants | 2.02 (0.15) | 1.96 (0.14) | 1.98 (0.18) | 1.93 (0.19) | 1.96 (0.11) | 1.97 (0.16)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 2.08 (0.12) | 1.93 (0.12) | 2.02 (0.15) | 1.96 (0.21) | 1.98 (0.09) | 1.99 (0.15)
Ultradistal tBV [Mean (Standard Deviation); unit: cm^3] — ultradistal endocortical bone volume measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  cm^3
    All Enrolled Participants | 1.47 (0.30) | 1.39 (0.23) | 1.41 (0.26) | 1.38 (0.31) | 1.42 (0.27) | 1.41 (0.27)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 1.55 (0.30) | 1.38 (0.24) | 1.45 (0.24) | 1.42 (0.32) | 1.46 (0.22) | 1.45 (0.26)
Ultradistal iBMD [Mean (Standard Deviation); unit: g/cm^3] — ultradistal integral volumetric bone mineral density measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g/cm^3
    All Enrolled Participants | 0.243 (0.044) | 0.238 (0.035) | 0.237 (0.030) | 0.228 (0.033) | 0.234 (0.031) | 0.236 (0.035)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.250 (0.044) | 0.230 (0.033) | 0.239 (0.032) | 0.233 (0.029) | 0.233 (0.029) | 0.237 (0.034)
Ultradistal cBMD [Mean (Standard Deviation); unit: g/cm^3] — ultradistal cortical volumetric bone mineral density measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g/cm^3
    All Enrolled Participants | 0.486 (0.035) | 0.471 (0.029) | 0.465 (0.028) | 0.473 (0.027) | 0.468 (0.014) | 0.473 (0.028)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.485 (0.039) | 0.469 (0.033) | 0.462 (0.029) | 0.470 (0.023) | 0.471 (0.013) | 0.471 (0.029)
Ultradistal ecBMD [Mean (Standard Deviation); unit: g/cm^3] — ultradistal endocortical volumetric bone mineral density measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g/cm^3
    All Enrolled Participants | 0.339 (0.097) | 0.307 (0.075) | 0.310 (0.067) | 0.289 (0.075) | 0.305 (0.059) | 0.310 (0.077)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.358 (0.092) | 0.286 (0.064) | 0.315 (0.080) | 0.301 (0.069) | 0.309 (0.063) | 0.312 (0.076)
Ultradistal tBMD [Mean (Standard Deviation); unit: g/cm^3] — ultradistal trabecular volumetric bone mineral density measured using quantitative computed tomography analysis of clinical resolution CT scans Population: All Enrolled Participants includes the 102 participants randomized into study arms. The Subset of Participants who were also Analyzed at Follow-up row reports baseline values for participants with 12 month follow-up data available, for more direct comparison with reported group changes.
  g/cm^3
    All Enrolled Participants | 0.122 (0.033) | 0.128 (0.031) | 0.129 (0.024) | 0.112 (0.031) | 0.127 (0.035) | 0.124 (0.031)
    Subset of Participants who were also Analyzed at Follow-Up (12 months): number analyzed (Participants) | 13 | 17 | 12 | 11 | 13 | 66
    Subset of Participants who were also Analyzed at Follow-Up (12 months) | 0.131 (0.022) | 0.121 (0.028) | 0.133 (0.027) | 0.120 (0.026) | 0.125 (0.033) | 0.126 (0.027)
Trabecular BV/TV [Mean (Standard Deviation); unit: ratio] — trabecular bone volume fraction expressed as the ratio of bone volume (BV) to total volume (TV) using: (BV/TV). This quantity is measured with high resolution peripheral quantitative computed tomography (HRpQCT). It is expressed as a ratio, ranging from 0 (none of the volume is occupied by bone) to 1 (all of the volume is occupied by bone). Population: Analysis population includes individuals with high quality baseline HRpQCT scans (motion artifact score <4).
  ratio
    number analyzed (Participants) | 18 | 23 | 21 | 20 | 15 | 97
    (all) | 0.131 (0.024) | 0.135 (0.026) | 0.138 (0.026) | 0.130 (0.024) | 0.141 (0.030) | 0.135 (0.026)
Cortical Thickness [Mean (Standard Deviation); unit: mm] — cortical thickness, measured with high resolution peripheral quantitative computed tomography (HRpQCT) Population: Analysis population includes individuals with high quality baseline HRpQCT scans (motion artifact score <4 according to Pialat et al. (2012) Bone).
  mm
    number analyzed (Participants) | 18 | 23 | 21 | 20 | 15 | 97
    (all) | 0.811 (0.168) | 0.753 (0.162) | 0.795 (0.154) | 0.828 (0.110) | 0.724 (0.085) | 0.784 (0.144)

OUTCOME MEASURES:

1. Primary Outcome: Change in UD iBMC
Description: 12-month change in ultra-distal integral bone mineral content, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g | 0.0049 (0.0146) | -0.0020 (0.0165) | 0.0252 (0.0206) | 0.0309 (0.0211) | -0.0106 (0.0241)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The power analysis for the overall study was based on 12-month change in UD iBMC. The power calculation, based on pilot data, determined that 20 participants per group would have 80% power to detect a 1.0±1.1% change. The null hypothesis was that change in UD iBMC was not proportional to strain magnitude. Raw change in iBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.119, Regression, Linear; Overall model fit: R^2=0.101, F=2.244, df1=2, df2=40, p=0.119 Contrast between the low strain magnitude group and the control group: B=0.015, Std. Error of estimate of B=0.007, Beta=0.374, t=2.114, p=0.041, 95% CI of B: [0.001, 0.030] Contrast between the high strain magnitude group and the control group: B=0.009, Std. Error of estimate of B=0.007, Beta=0.221, t=1.247, p=0.220, 95% CI of B: [-0.005, 0.022]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD iBMC was not proportional to strain rate. Raw change in iBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p < 0.01, Regression, Linear; Overall model fit: R^2=0.438, F=12.836, df1=2, df2=33, p=<0.001 Contrast between the low strain rate group and the control group: B=0.036, Std. Error of estimate of B=0.009, Beta=0.599, t=4.050, p=<0.001, 95% CI of B: [0.018, 0.055] Contrast between the high strain rate group and the control group: B=0.041, Std. Error of estimate of B=0.009, Beta=0.678, t=4.589, p=<0.001, 95% CI of B: [0.023, 0.060]

2. Secondary Outcome: Change in UD cBMC
Description: 12-month change in ultra-distal cortical bone mineral content, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g | 0.0037 (0.0127) | -0.0001 (0.0101) | 0.0139 (0.0124) | 0.0166 (0.0176) | 0.0024 (0.0243)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD cBMC was not proportional to strain magnitude. Raw change in cBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.809, Regression, Linear; Overall model fit: R^2=0.011, F=0.213, df1=2, df2=40, p=0.809 Contrast between the low strain magnitude group and the control group: B=0.001, Std. Error of estimate of B=0.006, Beta=0.039, t=0.209, p=0.836, 95% CI of B: [-0.012, 0.014] Contrast between the high strain magnitude group and the control group: B=-0.002, Std. Error of estimate of B=0.006, Beta=-0.077, t=-0.412, p=0.682, 95% CI of B: [-0.015, 0.010]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD cBMC was not proportional to strain rate. Raw change in cBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.155, Regression, Linear; Overall model fit: R^2=0.107, F=1.971, df1=2, df2=33, p=0.155 Contrast between the low strain rate group and the control group: B=0.012, Std. Error of estimate of B=0.008, Beta=0.284, t=1.526, p=0.137, 95% CI of B: [-0.004, 0.027] Contrast between the high strain rate group and the control group: B=0.014, Std. Error of estimate of B=0.008, Beta=0.342, t=1.837, p=0.075, 95% CI of B: [-0.002, 0.030]

3. Secondary Outcome: Change in UD ecBMC
Description: 12-month change in ultra-distal endocortical bone mineral content, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g | 0.0007 (0.0173) | 0.0001 (0.0151) | 0.0286 (0.0240) | 0.0287 (0.0274) | -0.0004 (0.0311)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD ecBMC was not proportional to strain magnitude. Raw change in ecBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.991, Regression, Linear; Overall model fit: R^2=<0.001, F=0.009, df1=2, df2=40, p=0.991 Contrast between the low strain magnitude group and the control group: B=0.001, Std. Error of estimate of B=0.009, Beta=0.025, t=0.133, p=0.894, 95% CI of B: [-0.016, 0.018] Contrast between the high strain magnitude group and the control group: B=0.001, Std. Error of estimate of B=0.008, Beta=0.012, t=0.063, p=0.950, 95% CI of B: [-0.016, 0.017]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD ecBMC was not proportional to strain rate. Raw change in ecBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.018, Regression, Linear; Overall model fit: R^2=0.216, F=4.548, df1=2, df2=33, p=0.018 Contrast between the low strain rate group and the control group: B=0.029, Std. Error of estimate of B=0.011, Beta=0.455, t=2.607, p=0.014, 95% CI of B: [0.006, 0.052] Contrast between the high strain rate group and the control group: B=0.029, Std. Error of estimate of B=0.011, Beta=0.447, t=2.563, p=0.015, 95% CI of B: [0.006, 0.052]

4. Secondary Outcome: Change in UD tBMC
Description: 12-month change in ultra-distal trabecular bone mineral content, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g | 0.0018 (0.0082) | -0.0021 (0.0067) | 0.0072 (0.0092) | 0.0112 (0.0106) | -0.0048 (0.0107)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD tBMC was not proportional to strain magnitude. Raw change in tBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.153, Regression, Linear; Overall model fit: R^2=0.090, F=1.968, df1=2, df2=40, p=0.153 Contrast between the low strain magnitude group and the control group: B=0.007, Std. Error of estimate of B=0.003, Beta=0.352, t=1.973, p=0.055, 95% CI of B: [0.000, 0.013] Contrast between the high strain magnitude group and the control group: B=0.003, Std. Error of estimate of B=0.003, Beta=0.156, t=0.874, p=0.387, 95% CI of B: [-0.004, 0.009]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD tBMC was not proportional to strain rate. Raw change in tBMC was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.001, Regression, Linear; Overall model fit: R^2=0.331, F=8.152, df1=2, df2=33, p=0.001 Contrast between the low strain rate group and the control group: B=0.012, Std. Error of estimate of B=0.004, Beta=0.473, t=2.930, p=0.006, 95% CI of B: [0.004, 0.020] Contrast between the high strain rate group and the control group: B=0.016, Std. Error of estimate of B=0.004, Beta=0.617, t=3.828, p=0.001, 95% CI of B: [0.008, 0.025]

5. Secondary Outcome: Change in UD iBMD
Description: 12-month change in ultra-distal integral volumetric bone mineral density, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g/cm^3 | -0.0008 (0.0024) | -0.0007 (0.0027) | 0.0072 (0.0027) | 0.0071 (0.0035) | -0.0014 (0.0047)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD iBMD was not proportional to strain magnitude. Raw change in iBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.840, Regression, Linear; Overall model fit: R^2=0.009, F=0.176, df1=2, df2=40, p=0.840 Contrast between the low strain magnitude group and the control group: B=0.001, Std. Error of estimate of B=0.001, Beta=0.091, t=0.489, p=0.628, 95% CI of B: [-0.002, 0.003] Contrast between the high strain magnitude group and the control group: B=0.001, Std. Error of estimate of B=0.001, Beta=0.101, t=0.544, p=0.589, 95% CI of B: [-0.002, 0.003]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD iBMD was not proportional to strain rate. Raw change in iBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p < 0.001, Regression, Linear; Overall model fit: R^2=0.563, F=21.225, df1=2, df2=33, p=<0.001 Contrast between the low strain rate group and the control group: B=0.009, Std. Error of estimate of B=0.002, Beta=0.739, t=5.669, p=<0.001, 95% CI of B: [0.005, 0.012] Contrast between the high strain rate group and the control group: B=0.008, Std. Error of estimate of B=0.002, Beta=0.716, t=5.495, p=<0.001, 95% CI of B: [0.005, 0.012]

6. Secondary Outcome: Change in UD cBMD
Description: 12-month change in ultra-distal cortical volumetric bone mineral density, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g/cm^3 | -0.0025 (0.0068) | -0.0015 (0.0073) | 0.0073 (0.0058) | 0.0036 (0.0081) | 0.0029 (0.0101)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD cBMD was not proportional to strain magnitude. Raw change in cBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.202, Regression, Linear; Overall model fit: R^2=0.077, F=1.665, df1=2, df2=40, p=0.202 Contrast between the low strain magnitude group and the control group: B=-0.005, Std. Error of estimate of B=0.003, Beta=-0.303, t=-1.689, p=0.099, 95% CI of B: [-0.012, 0.001] Contrast between the high strain magnitude group and the control group: B=-0.004, Std. Error of estimate of B=0.003, Beta=-0.266, t=-1.484, p=0.146, 95% CI of B: [-0.010, 0.002]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD cBMD was not proportional to strain rate. Raw change in cBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.381, Regression, Linear; Overall model fit: R^2=0.057, F=0.995, df1=2, df2=33, p=0.381 Contrast between the low strain rate group and the control group: B=0.004, Std. Error of estimate of B=0.003, Beta=0.254, t=1.327, p=0.194, 95% CI of B: [-0.002, 0.011] Contrast between the high strain rate group and the control group: B=0.001, Std. Error of estimate of B=0.003, Beta=0.038, t=0.200, p=0.843, 95% CI of B: [-0.006, 0.008]

7. Secondary Outcome: Change in UD ecBMD
Description: 12-month change in ultra-distal endocortical bone mineral density, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g/cm^3 | -0.0031 (0.0102) | -0.0012 (0.0080) | 0.0141 (0.0105) | 0.0122 (0.0116) | 0.0005 (0.0141)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD ecBMD was not proportional to strain magnitude. Raw change in ecBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.697, Regression, Linear; Overall model fit: R^2=0.018, F=0.365, df1=2, df2=40, p=0.697 Contrast between the low strain magnitude group and the control group: B=-0.004, Std. Error of estimate of B=0.004, Beta=-0.158, t=-0.854, p=0.398, 95% CI of B: [-0.012, 0.005] Contrast between the high strain magnitude group and the control group: B=-0.002, Std. Error of estimate of B=0.004, Beta=-0.078, t=-0.423, p=0.675, 95% CI of B: [-0.010, 0.006]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD ecBMD was not proportional to strain rate. Raw change in ecBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.018, Regression, Linear; Overall model fit: R^2=0.215, F=4.516, df1=2, df2=33, p=0.018 Contrast between the low strain rate group and the control group: B=0.014, Std. Error of estimate of B=0.005, Beta=0.484, t=2.773, p=0.009, 95% CI of B: [0.004, 0.0524] Contrast between the high strain rate group and the control group: B=0.012, Std. Error of estimate of B=0.005, Beta=0.406, t=2.325, p=0.026, 95% CI of B: [0.001, 0.022]

8. Secondary Outcome: Change in UD tBMD
Description: 12-month change in ultra-distal trabecular bone mineral density, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
g/cm^3 | 0.0006 (0.0028) | -0.0013 (0.0036) | 0.0050 (0.0043) | 0.0071 (0.0053) | -0.0029 (0.0046)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD tBMD was not proportional to strain magnitude. Raw change in tBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.073, Regression, Linear; Overall model fit: R^2=0.123, F=2.799, df1=2, df2=40, p=0.073 Contrast between the low strain magnitude group and the control group: B=0.003, Std. Error of estimate of B=0.001, Beta=0.413, t=2.361, p=0.023, 95% CI of B: [0.000, 0.006] Contrast between the high strain magnitude group and the control group: B=0.002, Std. Error of estimate of B=0.001, Beta=0.198, t=1.129, p=0.265, 95% CI of B: [-0.001, 0.004]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD tBMD was not proportional to strain rate. Raw change in tBMD was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p < 0.001, Regression, Linear; Overall model fit: R^2=0.480, F=15.256, df1=2, df2=33, p=<0.001 Contrast between the low strain rate group and the control group: B=0.008, Std. Error of estimate of B=0.002, Beta=0.590, t=4.153, p=<0.001, 95% CI of B: [0.004, 0.012] Contrast between the high strain rate group and the control group: B=0.001, Std. Error of estimate of B=0.002, Beta=0.734, t=5.164, p=<0.001, 95% CI of B: [0.006, 0.014]

9. Secondary Outcome: Change in UD iBV
Description: 12-month change in ultra-distal integral bone volume, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
cm^3 | 0.027 (0.061) | 0.003 (0.055) | -0.011 (0.049) | 0.012 (0.066) | -0.026 (0.068)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD iBV was not proportional to strain magnitude. Raw change in iBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.101, Regression, Linear; Overall model fit: R^2=0.108, F=2.428, df1=2, df2=40, p=0.101 Contrast between the low strain magnitude group and the control group: B=0.053, Std. Error of estimate of B=0.024, Beta=0.388, t=2.200, p=0.034, 95% CI of B: [0.004, 0.101] Contrast between the high strain magnitude group and the control group: B=0.029, Std. Error of estimate of B=0.022, Beta=0.226, t=1.280, p=0.208, 95% CI of B: [-0.017, 0.074]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD iBV was not proportional to strain rate. Raw change in iBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.344, Regression, Linear; Overall model fit: R^2=0.063, F=01.103, df1=2, df2=33, p=0.344 Contrast between the low strain rate group and the control group: B=0.015, Std. Error of estimate of B=0.025, Beta=0.113, t=0.595, p=0.556, 95% CI of B: [-0.036, 0.065] Contrast between the high strain rate group and the control group: B=0.038, Std. Error of estimate of B=0.025, Beta=0.283, t=1.481, p=0.148, 95% CI of B: [-0.014, 0.089]

10. Secondary Outcome: Change in UD cBV
Description: 12-month change in ultra-distal cortical bone volume, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
cm^3 | 0.014 (0.028) | 0.003 (0.028) | 0.016 (0.035) | 0.031 (0.038) | 0.002 (0.056)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD cBV was not proportional to strain magnitude. Raw change in cBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.676, Regression, Linear; Overall model fit: R^2=0.019, F=0.395, df1=2, df2=40, p=0.676 Contrast between the low strain magnitude group and the control group: B=0.012, Std. Error of estimate of B=0.015, Beta=0.146, t=0.787, p=0.436, 95% CI of B: [-0.019, 0.042] Contrast between the high strain magnitude group and the control group: B=0.001, Std. Error of estimate of B=0.014, Beta=0.013, t=0.070, p=0.945, 95% CI of B: [-0.028, 0.029]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD cBV was not proportional to strain rate. Raw change in cBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.289, Regression, Linear; Overall model fit: R^2=0.072, F=1.288, df1=2, df2=33, p=0.289 Contrast between the low strain rate group and the control group: B=0.014, Std. Error of estimate of B=0.018, Beta=0.154, t=0.814, p=0.422, 95% CI of B: [-0.022, 0.051] Contrast between the high strain rate group and the control group: B=0.029, Std. Error of estimate of B=0.018, Beta=0.304, t=1.604, p=0.118, 95% CI of B: [-0.008, 0.066]

11. Secondary Outcome: Change in UD ecBV
Description: 12-month change in ultra-distal cortical bone volume, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
cm^3 | 0.018 (0.029) | 0.008 (0.030) | -0.0003 (0.025) | 0.009 (0.028) | -0.007 (0.030)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD ecBV was not proportional to strain magnitude. Raw change in ecBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.096, Regression, Linear; Overall model fit: R^2=0.111, F=2.491, df1=2, df2=40, p=0.096 Contrast between the low strain magnitude group and the control group: B=0.026, Std. Error of estimate of B=0.012, Beta=0.391, t=2.222, p=0.032, 95% CI of B: [0.032, 0.049] Contrast between the high strain magnitude group and the control group: B=0.015, Std. Error of estimate of B=0.011, Beta=0.240, t=1.362, p=0.181, 95% CI of B: [-0.007, 0.037]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD ecBV was not proportional to strain rate. Raw change in ecBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.344, Regression, Linear; Overall model fit: R^2=0.063, F=1.103, df1=2, df2=33, p=0.344 Contrast between the low strain rate group and the control group: B=0.014, Std. Error of estimate of B=0.015, Beta=0.113, t=0.595, p=0.556, 95% CI of B: [-0.036, 0.065] Contrast between the high strain rate group and the control group: B=0.038, Std. Error of estimate of B=0.025, Beta=0.283, t=1.481, p=0.148, 95% CI of B: [-0.014, 0.089]

12. Secondary Outcome: Change in UD tBV
Description: 12-month change in ultra-distal trabecular bone volume, measured with quantitative computed tomography (QCT)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 13 | 17 | 12 | 11 | 13
cm^3 | 0.006 (0.029) | -0.004 (0.023) | -0.003 (0.023) | 0.006 (0.034) | -0.011 (0.033)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in UD tBV was not proportional to strain magnitude. Raw change in tBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.332, Regression, Linear; Overall model fit: R^2=0.054, F=1.132, df1=2, df2=40, p=0.332 Contrast between the low strain magnitude group and the control group: B=0.016, Std. Error of estimate of B=0.011, Beta=0.271, t=1.493, p=0.143, 95% CI of B: [-0.006, 0.039] Contrast between the high strain magnitude group and the control group: B=0.007, Std. Error of estimate of B=0.010, Beta=0.115, t=635, p=0.529, 95% CI of B: [-0.014, 0.028]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in UD tBV was not proportional to strain rate. Raw change in tBV was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p = 0.399, Regression, Linear; Overall model fit: R^2=0.054, F=0.946, df1=2, df2=33, p=0.399 Contrast between the low strain rate group and the control group: B=0.008, Std. Error of estimate of B=0.012, Beta=0.119, t=0.619, p=0.540, 95% CI of B: [-0.017, 0.032] Contrast between the high strain rate group and the control group: B=0.017, Std. Error of estimate of B=0.012, Beta=0.264, t=1.375, p=0.178, 95% CI of B: [-0.008, 0.042]

13. Secondary Outcome: Change in Cortical Thickness
Description: Changes in cortical thickness at 3-month intervals, measured with high resolution peripheral quantitative computed tomography (HRpQCT)
Time Frame: measurements repeated at 0, 3, 6, 9, 12, 18, and 24 months from enrollment
Population: Analysis population includes participants analyzed at at least one interim timepoint. Exact values are provided for individual timepoints below.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 15 | 21 | 15 | 11 | 15
mm
  3 months: number analyzed (Participants) | 9 | 18 | 9 | 10 | 10
  3 months | 0.001 (0.018) | -0.012 (0.056) | 0.009 (0.030) | 0.032 (0.031) | -0.004 (0.018)
  6 months: number analyzed (Participants) | 13 | 14 | 11 | 10 | 14
  6 months | -0.003 (0.037) | 0.002 (0.021) | 0.008 (0.025) | 0.005 (0.025) | 0.004 (0.018)
  9 months: number analyzed (Participants) | 11 | 12 | 12 | 7 | 12
  9 months | 0.001 (0.015) | -0.012 (0.064) | 0.006 (0.019) | -0.007 (0.022) | -0.002 (0.021)
  12 months: number analyzed (Participants) | 12 | 14 | 11 | 9 | 11
  12 months | -0.009 (0.027) | -0.002 (0.027) | 0.015 (0.018) | 0.004 (0.029) | 0.002 (0.022)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in cortical thickness was not proportional to strain magnitude. At each time point, raw change relative to baseline was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; At each time point, the overall fit of the linear regression model was assessed with an F-test of overall significance. Additionally, the significance of each coefficient representing contrasts between each experimental group and the control group was assessed using t-tests. There were no significant relationships found between change in cortical thickness and strain magnitude group at any time point (p>0.05)
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in cortical thickness was not proportional to strain rate. At each time point, raw change relative to baseline was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; At each time point, the overall fit of the linear regression model was assessed with an F-test of overall significance. Additionally, the significance of each coefficient representing contrasts between each experimental group and the control group was assessed using t-tests. At 3 months, there was a significant overall linear relationship between change in cortical thickness and strain rate group. Additionally, the coefficient representing the contrast between the control group and the high strain rate group was also significant. All other comparisons were not statistically significant (p>0.05). Stats for 3 months: Overall model fit: R^2=0.258, F=4.519, df1=2, df2=26, p=0.021 Contrast between the high strain rate group and the control group: B=0.036, Std. Error of estimate of B=0.012, Beta=0.574, t=2.967, p=0.006, 95% CI of B: [0.011, 0.061]

14. Secondary Outcome: Change in Trabecular BV/TV
Description: trabecular bone volume fraction expressed as the ratio of bone volume (BV) to total volume (TV) using: (BV/TV). This quantity is measured with high resolution peripheral quantitative computed tomography (HRpQCT). It is expressed as a ratio, ranging from 0 (none of the volume is occupied by bone) to 1 (all of the volume is occupied by bone).
Time Frame: measurements repeated at 0, 3, 6, 9, and 12 months from enrollment
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
Number analyzed (Participants) | 15 | 21 | 15 | 11 | 15
ratio
  3 months: number analyzed (Participants) | 9 | 18 | 9 | 10 | 10
  3 months | -0.0006 (0.0023) | 0.0003 (0.0030) | -0.0020 (0.0044) | 0.0002 (0.0025) | -0.0014 (0.0021)
  6 months: number analyzed (Participants) | 13 | 14 | 11 | 10 | 14
  6 months | 0.0006 (0.0030) | -0.0004 (0.0031) | 0.0011 (0.0027) | 0.0008 (0.0030) | -0.0007 (0.0032)
  9 months: number analyzed (Participants) | 11 | 12 | 12 | 7 | 12
  9 months | 0.0014 (0.0020) | -0.0004 (0.0027) | 0.0003 (0.0030) | -0.0001 (0.0034) | -0.0020 (0.0028)
  12 months: number analyzed (Participants) | 12 | 14 | 11 | 9 | 11
  12 months | 0.0002 (0.0026) | 0.0010 (0.0033) | 0.0009 (0.0032) | 0.0007 (0.0034) | 0.000 (0.0048)
Statistical Analysis 1: Comparison: Low Magnitude vs High Magnitude vs Control; The null hypothesis was that change in bone volume fraction (BV/TV) was not proportional to strain magnitude. At each time point, raw change relative to baseline was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; At each time point, the overall fit of the linear regression model was assessed with an F-test of overall significance. Additionally, the significance of each coefficient representing contrasts between each experimental group and the control group was assessed using t-tests. At 9 months, there was a significant overall linear relationship between change in BV/TV and strain magnitude group. Additionally, the coefficient representing the contrast between the control group and the low strain magnitude group was also significant. All other comparisons were not statistically significant (p>0.05). Stats for 9 months: Overall model fit: R^2=0.240, F=5.057, df1=2, df2=32, p=0.012 Contrast between the low strain magnitude group and the control group: B=0.003, Std. Error of estimate of B=0.001, Beta=0.562, t=3.180, p=0.003, 95% CI of B: [0.001, 0.006]
Statistical Analysis 2: Comparison: Low Rate vs High Rate vs Control; The null hypothesis was that change in bone volume fraction (BV/TV) was not proportional to strain rate. At each time point, raw change relative to baseline was analyzed as the dependent variable in a linear regression model with coefficients representing contrasts between the two experimental groups and the control group; Test type: Other; p > 0.05, Regression, Linear; At each time point, the overall fit of the linear regression model was assessed with an F-test of overall significance. Additionally, the significance of each coefficient representing contrasts between each experimental group and the control group was assessed using t-tests

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant for the 2-year study period following enrollment.
Description: At each visit, the standard Study Visit Data Collection Sheet recorded whether participants had experienced in the past 3 months:
  1. Aches or pain in the non-dominant wrist
  2. Fractures
  3. Other problems that you think might be associated with participating in this research
  4. Other problems that have prevented you from completing your assigned intervention
Arm/Group | Low Magnitude | High Magnitude | Low Rate | High Rate | Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/24 | 0/21 | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24 | 0/21 | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 8/21 | 11/24 | 10/21 | 11/20 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Magnitude (N=21) | High Magnitude (N=24) | Low Rate (N=21) | High Rate (N=20) | Control (N=16)
Temporary Wrist Soreness (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6) | 8 (11) | 8 (10) | 3 (4) — Includes wrist soreness, potentially related to the intervention for exercise participants. Also includes other causes of wrist soreness such as overuse injury, sprain, and carpal tunnel for intervention and control groups.
Arm Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 3 (5) | 2 (2) — Elbow, shoulder, or hand pain, potentially related to the intervention or not related to the intervention. Includes several cases of aggravation of previous injuries potentially due to the intervention.
Other injury or pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) — Includes back and lower limb injuries not related to the intervention reported by participants in the load and control groups.
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant experienced anxiety during blood draw during the initial screening visit.
Wrist Bump (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported bump on wrist potentially related to the intervention. The bump went away 3 months after discontinuing the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT04135196/Prot_001.pdf
  • Statistical Analysis Plan (2012-01-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04135196/SAP_002.pdf
  • Informed Consent Form (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04135196/ICF_003.pdf